CLINICAL TRIAL: NCT06308211
Title: Comparative Effects of Motor Imagery and Mirror Therapy Versus Motor Relearning Program on Balance, Motor Function and Activities of Daily Living in Subacute Stroke Patients
Brief Title: Comparative Effects of Motor Imagery and Mirror Therapy Versus Motor Relearning Program in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0289
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Mirror therapy; Motor relearning Programme; stroke; Motor Imagery
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient would be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (MOTOR IMAGERY+MIRROR THERAPY+ROUTINE PHYSICAL THERAPY) (Experimental): Group A will receive treatment session of 60 minutes including motor imagery for 20 minutes and mirror therapy for 20 minutes along with routine physical therapy of 20 minutes for 5 days per week for 12 weeks.In motor imagery subjects will watch the video and will be asked to close the eyes to focus and imagine how they are doing task they had previously observed 10 times and instructed to carry out the task in verbal commands given whenever necessary.
  In mirror therapy,The unaffected limb will be placed in front of the mirror and patient will try to make the identical motions with the paretic limb while moving the non-paretic limb during the session and routine physical therapy includes passive and active assisted range of motion for the upper and lower extremity including the shoulder, forearm, wrist, hip, knee and ankle will be given (10 - 15 repititions).
  Interventions: Other: MOTOR IMAGERY+MIRROR THERAPY+ROUTINE PHYSICAL THERAPY
- GROUP B (MOTOR RELEARNING PROGRAM+ROUTINE PHYSICAL THERAPY) (Experimental): GROUP B will receive treatment session of 60 minutes including motor relearning program of 40 minutes duration along with routine physical therapy of 20 minutes as explained in group A protocol. Treatment session will be given 5 days per week for 12 weeks.
  Motor relearning consists of five components including analysis of task, practice of missing components, practice of task and transference of training.
  Interventions: Other: MOTOR RELEARNING PROGRAM+ROUTINE PHYSICAL THERAPY

INTERVENTIONS:
Other: MOTOR IMAGERY+MIRROR THERAPY+ROUTINE PHYSICAL THERAPY — Subjects will be instructed to watch the video provided and recorded by investigator.In next step participants will be asked to close the eyes to focus and then to imagine how they are doing task they had previously observed 10 times.Participants will be than instructed to carry out the task in verbal commands given whenever necessary.The unaffected limb will be placed in front of the mirror so that the reflected illusion of the limb would be hallucinated to represent the affected limb and routine physical therapy includes passive and active assisted range of motion for the upper and lower extremity including the shoulder, forearm, wrist, hip, knee and ankle will be given (10 - 15 repititions).
  Other Names: Rehabilitation
  Arms: GROUP A (MOTOR IMAGERY+MIRROR THERAPY+ROUTINE PHYSICAL THERAPY)
Other: MOTOR RELEARNING PROGRAM+ROUTINE PHYSICAL THERAPY — Motor relearning consists of five components including analysis of task, practice of missing components, practice of task and transference of training. Patient will be asked to practice task in both sitting and standing
  * supine to side-lying to sitting
  * looking up at ceiling (ensure that centre of body mass does not move back when head is tilted back)
  * without moving one's feet, turning to gaze over each other's shoulders and scanning the surroundings for specific items, reaching motions in multiple directions while moving the head and trunk, scooting in bed, altering the base of support (standing with your feet together, in tandem, with one foot on a step, or on one leg)
  * squatting to pick up an object and cross over stepping and routine physical therapy includes Passive and active assisted range of motion for the upper and lower extremity including the shoulder, forearm, wrist, hip, knee and ankle will be given (10 - 15 repititions).
  Other Names: Rehabilitation
  Arms: GROUP B (MOTOR RELEARNING PROGRAM+ROUTINE PHYSICAL THERAPY)

SUMMARY:
Use of motor imagery, mirror therapy and motor relearning program in rehabilitation of people with stroke is on rise and these are unique and emerging techniques. Motor imagery is a mental rehearsal through visualization while mirror therapy creates a reflection of non-effected limb by using a mirror. Moreover, motor relearning is task-oriented approach, benefacial for balance and motor funCtion in patients with stroke that emphasizes on relearning.The aim of the study is to determine the comparative effects of motor imagery and mirror therapy versus motor relearning program in addition to routine physical therapy on balance, motor function and activities of daily living in subacute stroke patients.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at medical centre Fifty stroke patients will be included using convenience sampling technique. The participants in the study will be randomly allocated in to two groups . Twenty five participants will be included in both Groups A d B. Group A (motor imagery and mirror therapy) will receive 60 minutes treatment session that consists of 20 minutes motor imagery, 20 minutes mirror therapy along with 20 minutes routine physical therapy and Group B (motor relearning program) will receive treatment session of 60 minutes including motor relearning program of 40 minutes duration along with routine physical therapy of 20 minutes. Both groups will undergo 60 minutes session for 5 days per week for 12 weeks. Berg balance scale will be used to assess balance, Fugl-meyer assessment to assess motor function and Functional independence measure for activities of daily living. Assessment will be carried out at baseline, 4th week, 8th week and at 12th week after the discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke patient of both gender.
2. Stroke patient of age 40-65 year .
3. Patient diagnosis of cerebral ischemic stroke .
4. Patients who had suffered a stroke with hemiplegia, were subacute at least 3 months to 5 months since the onset.
5. Ability to walk with minimal assistance (functional ambulation category 1 to 3.
6. Patient with score > 25 on mini-mental status examination.

Exclusion Criteria:

1. Patients who presented with hemiplegic neglect or apraxia
2. Patients with history of global or receptive aphasia
3. Patients with history of psychological or emotional problems
4. Patients with history of decompensated cardiovascular/ respiratory/ digestive/ renal disorders, biologic inflammatory syndrome, neoplastic disorders, neurogenic bladder or skin disorders (bedsores).
5. Patients with history of artificial joints

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Berg balance scale (BBS) | 12th week
  The BBS is postural balance scale containing 14 items including standing and sitting unsupported, reaching forward, and placing the alternating foot on a stool. Administering the BBS takes approximately 15 min. Each of the 14 items are scored on a 5-level ordinal scale from 0 ("unable to perform or requiring help") to 4 ("normal performance"), thus providing a potential maximum score of 56 points
FUGL-MEYER ASSESMENT (FMA) | 12th week
  The Fugl-Meyer Assessment is a welldesigned, feasible and efficient clinical examination method that has been tested widely in the stroke population. A three-level ordinal scale (0, can perform no part of the test; 1, performs test partially; 2, performs test normally) is applied to each item. A total possible score for the lower extremity is 34. The higher the score, the better the performance.
FUNCTIONAL INDEPENDENCE MEASURE (FIM) | 12th week
  The Functional Independence Measure (FIM) is one of the most frequently used outcome measures in stroke rehabilitation trials. The five FIM items dealing with transfers and locomotion, including transfers to bed/chair/wheelchair, toileting, bathing, walking or wheelchair management and stairs, were used in this pilot study to evaluate the activities of daily living in the patients with stroke. Each item is rated on a seven-level scale, with 1 = total assistance and 7 (complete independence). By adding the points for each item in the transfers and locomotion, the possible total score ranges from 5 (lowest) to 35 (highest) level of independence; the higher the score, the better the independence. This scale has good reliability for the assessment of recovery of function in stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD, Study Chair — Riphah International University
Locations (1):
- Muhammad Kashif, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No